CLINICAL TRIAL: NCT03165656
Title: Right Ventricular Function at Rest in Highlanders With Pulmonary Hypertension Compared to Highlanders Without Pulmonary Hypertension and Lowlanders
Brief Title: Right Ventricular Function at Rest in Highlanders/Lowlanders
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Principal Investigator, Silvia Ulrich Somaini, Prof. Dr., University of Zurich
Other Study IDs: 01-8/433A
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Echocardiography; right ventricular function; pulmonary hypertension; disease progression; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Disease Progression; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High altitude pulmonary hypertension: Highlanders with high altitude pulmonary hypertension living above 2500 m.
- High altitude control: Healthy highlanders living above 2500 m.
- Low altitude control: Healthy lowlanders living below 1000 m.

SUMMARY:
The purpose of the current study is to evaluate the progression of right ventricular function and dimension in Kyrgyz highlanders with high altitude pulmonary hypertension (HAPH) by performing a cross sectional case-control study.

ELIGIBILITY:
Inclusion Criteria:

* high altitude pulmonary hypertension confirmed by clinical presentation and mean pulmonary artery pressure >30 mmHg measured by echocardiography at altitude of residence.
* healthy subjects (high altitude controls)
* Both genders
* Age >16 y
* Kyrgyz ethnicity
* born, raised and currently living at >2500 m
* healthy subjects currently living at <1000 m (low altitude controls)

Exclusion Criteria:

* Pulmonary hypertension from other causes, in particular from left ventricular failure as judged clinically and by echocardiography
* Excessive erythrocytosis
* Other coexistent disorders that may interfere with the cardio-respiratory system and sleep
* Regular use of medication that affects control of breathing
* Heavy smoking

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Highlanders with high altitude pulmonary hypertension living at an altitude of 2500-4000 m; healthy highlanders living at an altitude of 2500-4000 m; healthy lowlanders living at an altitude of <1000 m.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery pressure | Day 2
  Difference between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders in tricuspid pressure gradient, measured by transthoracic echocardiography

SECONDARY OUTCOMES:
cardiac output | Day 2
  Difference between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders in cardiac output, measured by transthoracic echocardiography
right heart dimensions | Day 2
  Difference of right heart dimensions between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography
Right heart function | Day 2
  Differences of right heart function between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography (TAPSE)
stroke volume | Day 2
  Difference between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders in stroke volume, measured by transthoracic echocardiography
volumes | Day 2
  Difference of volumes between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, MD, Study Chair — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gosens R, Hiemstra PS, Adcock IM, Bracke KR, Dickson RP, Hansbro PM, Krauss-Etschmann S, Smits HH, Stassen FRM, Bartel S. Host-microbe cross-talk in the lung microenvironment: implications for understanding and treating chronic lung disease. Eur Respir J. 2020 Aug 20;56(2):1902320. doi: 10.1183/13993003.02320-2019. Print 2020 Aug. PMID 32430415